CLINICAL TRIAL: NCT03406845
Title: Brief Chair-Side Mindfulness Intervention for Depression and Anxiety Symptoms in Patients Undergoing Dialysis: A Pilot Randomized Control Trial With an Active Control Group
Brief Title: Mindfulness and HEP in Dialysis Patients With Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); University of Toronto (Other); University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Soham Rej MD, MSc, Psychiatris and researcher, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MM-CODIM-MBM-17-169
Record Dates: First submitted 2017-11-29; First posted 2018-01-23 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Renal Disease; Depression; Anxiety
MeSH Terms: conditions — Kidney Diseases; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Masking Description: As described above.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chair-side mindfulness intervention (Experimental): Consists of individually conducted meditative practices, lasting 20 minutes/session, 3 times per week for 8 weeks. The interventions will be conducted during their dialysis sessions. The mindfulness meditation sessions include well-described meditations such as the body scan (being aware of bodily sensation), gentle arm movements, guided and silent breath meditations.
  Interventions: Behavioral: Chair-side mindfulness intervention
- Health Enhancement Plan (HEP) (Active Comparator): Has been previously designed and used for the purpose of being a manualized active control in meditation-based intervention trials, controlling for several non-specific factors found in a mindfulness meditation group. Participants will learn about health promotion, healthy diet, music, exercise as well as implementing positive health-enhancing life changes both in-session and during at-home practice with the support of a group facilitator, but do not learn mindfulness techniques.
  Interventions: Behavioral: Chair-side mindfulness intervention

INTERVENTIONS:
Behavioral: Chair-side mindfulness intervention — Tailored mindfulness intervention to chair-side type, based from Mindfulness Based Cognitive Therapy (MBCT).
  Health promotion based on the Health Enhancement Program (HEP).
  Other Names: HEP active control

SUMMARY:
This pilot clinical trial examines the acceptability of meditation techniques versus health promotion in people receiving dialysis who have anxiety or depression. 50% of people who undergo dialysis experience anxiety or depression, but these conditions go undetected and untreated. Meditation and help promotion is helpful for anxiety and depression, but no one has compared the effects of meditation versus health promotion in people on dialysis specifically. Our aim is to evaluate whether meditation is more effective than health promotion.

Nephrology doctors and nurses from collaborating hospitals in Montreal (MUHC) will help the recruit participants. The study will last 8 weeks, including a 6-month follow-up to measure depression and anxiety symptoms. Assessment will include pre-post evaluations about their depression and anxiety symptoms, overall health, sleep (Acti-watch), heart rate variability and blood draws (for inflammatory markers). A qualitative interview assessing participant experience will take place at program end.

Participants will be randomly assigned. The participants will practice meditation or health promotion exercises with a trained interventionist in 20-minute sessions 3 times a week, during their dialysis sessions. Participants in the meditation group will learn mindfulness meditation exercises, whereas participants in the health promotion group will learn about healthy diet, music, exercise and positive health-enhancing life changes.

Many people find meditation and health promotion enjoyable and relaxing. In the unlikely event people may have intense, but not dangerous reactions to meditation, the interventionists are trained to manage their reaction and direct them to appropriate care. Their hemodialysis treatment will not be affected by this study.

It is hoped to improve mental health care for people on dialysis suffering from depression and anxiety. If this study shows that people in the meditation group greatly benefited than those participating in health promotion, investigators will create a bigger study to confirm whether it is truly effective for anxiety and depression in dialysis patients. Meditation may become a widely used treatment for people on dialysis with anxiety and depression, and investigators would train nephrology staff to make this treatment as accessible as possible.

DETAILED DESCRIPTION:
Background Dialysis patients are prone to lower increased non-adherence, suicidal behavior, medical comorbidity, mortality and low quality of life. As a result of illness burden in dialysis, treatment is costly and resources for treatment allocation are on the rise. In the United States alone, costs per year of dialysis are US$67,000 for Medicare patients and US$80,000 for employer group health plan patients, and the worldwide consensus on estimates for total therapy cost in dialysis indicate that hospital dialysis is more expensive that non-hospital dialysis. Moreover, depression and anxiety are highly costly to health systems and society, and are the most common mental health symptoms in patients on maintenance dialysis (e.g. 50% of patients experience depression and anxiety symptoms) as supported by our recent cross-sectional study of 80 dialysis patients in Toronto and Montreal. Additionally, estimates of depression and anxiety diagnoses based on psychiatric interview in patients in dialysis vary between 20% and 30%, classifying depression as most common in patients on dialysis compared to the regular population.

Patients' views on dialysis treatment: treatment adherence and health outcomes. Limited studies investigating dialysis views convey barriers to adherence to pharmacological treatment, including doubts about the effectiveness of medications, complicated healthcare systems, and financial difficulties. This is significant, given patients need to have a sense of control, demonstrate self-efficacy and trust the advice from health care providers for shared decision-making and to maintain quality of life. Moreover, special attention has been paid to the study of patient perspectives in depression and anxiety, especially as important barriers to treatment retention include symptomatology display. In dialysis patients, depression plays an important role in adherence of treatment as patient report insufficient counselling and support during treatment; the high proportion of multiple disabilities experienced during treatment inevitably decreases patient's quality of life and augments outcomes related to poor health (e.g. insomnia). It is therefore important to study illness and health perceptions on treatment outcome as these may not only serve to improve adherence of dialysis treatment, but other health outcomes.

Limitations of existing treatments for depression and anxiety in dialysis patients. Given that depression and anxiety are associated with lower quality of life, disability, mortality, increased hospitalizations, shortened survival, increased dialysis non-adherence and suicidal behavior, dialysis patients' themselves have identified depression and anxiety as priorities for treatment and research. Existing health service delivery approaches, such as use of psychotropic medication and psychotherapy have been inadequate, resource-intensive, and are not financially feasible. First, there is often little interest from users and providers to modify or use antidepressant treatment as an effort to improve depression management. Current reports reiterating the issue of recruitment to antidepressant trials have identified concerns to pill burden (e.g. antidepressant dependency and increased side-effects), large dropout rates and low adherence to medication. Second, the role of competing factors (e.g. high symptom burden, inter-current events, and kidney disease-related losses) challenge the interpretation of results from trials conducted to depression treatment in dialysis and non prioritizing its treatment. Third, time requirements of dialysis treatment, patient tiredness before and after treatment, are impractical to patients' compliance to participate in psychosocial interventions. Also, there is no clear evidence to use Cognitive Behavioral Therapy (CBT) as a mean to alleviate symptoms of depression. This is of particular concern in the attempt to implement feasible and sustainable interventions in clinical practice, given the small number of studies reporting patient consent rates and uptake to these types of interventions.

Mindfulness-based interventions for dialysis patients. New "third" wave therapies including mindfulness-based interventions have gained increasing popularity in recent years as approaches to reduce psychological morbidity and emotional distress in physical and mental illness. Mindfulness involves learning concentration and relaxation techniques that allow practitioners to enter into present-moment awareness where the mind is simultaneously focused and relaxed. Such relaxed, yet focused mental states can help with depression and anxiety by teaching patients to be in the present moment, reducing the impact of negative cognitions and self-judgemental thoughts that often occur in anxiety and depression. Mindfulness-based Cognitive Therapy (MBCT) has been highly effective in treating chronic physical illness and many other conditions, including cancer. To our knowledge, literature reports on mindfulness for the treatment of depression hemodialysis are very limited. Some researchers have examined the effect of mindfulness-based psychotherapy and acceptance and commitment therapy on dialysis patients, but our group has been the first to explore the feasibility of brief chair-side mindfulness meditation for depression and anxiety symptoms in patients undergoing dialysis.

Preliminary results- Brief mindfulness intervention for patients undergoing hemodialysis. This group of researchers have completed a pilot randomized controlled trial (RCT) comparing brief mindfulness meditation (n=21) to treatment-as-usual (n=30), where the intervention was found feasible and enjoyable for patients on dialysis despite several systemic barriers. Of the participants randomized to the intervention group, 71% completed the study, with meditation being well-tolerated (median rating of 8/10 in Likert scale). Meditation was associated with subjective benefits but no significant impact on depression scores (change in PHQ9 -3.00±3.93 in the intervention group vs. - 2.00±4.74 in controls, p=0.45) or anxiety scores (change in GAD-7 -0.94±4.59 vs. -0.80±4.84, p=0.91). In this pilot sample, the intervention did not have statistically significant effects on depression and anxiety symptoms, except in a subgroup with more impairing baseline symptom, where it was beneficial (clinically important reduction in depressive symptom scores -4.29±3.5 vs. +0.14±3.5, p=0.034, n=14, 34% of sample).

Our findings suggested that although a chair-side mindfulness intervention is appreciated by dialysis patients, a number of modifications could improve impact: targeting patients with more significant baseline depressive or anxiety symptoms, incorporating a cognitive therapy component to better understand how to apply mindfulness in daily life, and finding novel ways to improve scalability. The next step is a pilot RCT with an active control group controlling for clinical attention and support to estimate the sample size of a definitive RCT. Investigators propose to strengthen our experimental design by addressing sustained treatment effects of chair-side mindfulness intervention while compared to the Health Enhancement Program (HEP)- a validated active control.

Inflammatory response in dialysis patients. Patients undergoing dialysis also often have a high burden of systemic inflammation, including elevated blood inflammation biomarkers. This in turn triggers a cascade that has been extensively shown in humans and animals to cause depressive symptoms, due to the permeability of blood endothelial cells, followed by activation of inflammatory pathways in the brain (28442354) and consequently, symptoms of depression. A possible association between these pro-inflammatory cytokines and the symptoms of depression can better explain the high rates of depression and the non-adherence to treatment in patients undergoing dialysis. Recent evidence suggests that mind-body therapies decrease the levels of the inflammation biomarkers such as inflammatory transcription factor NFKB (nuclear factor kB), which also has been associated with lower symptoms of anxiety and depression. Thus, an association between these two components can better explain the high rates of depression, non-adherence to treatment and can be a predictor of poor antidepressant and psychotherapy response. Therefore, it may be of great interest to explore whether inflammation is a predictor of depression/anxiety response in dialysis patients and whether mindfulness can improve inflammation in dialysis patients.

To circumvent the urge to improve the lives of patients with kidney disease in the near term and with widespread applicability, our group suggests the use of a brief chair-side mindfulness intervention as a compelling treatment adjunct to alleviate symptoms of depression and anxiety using a validated active control (HEP). This study will also investigate whether brief chair-side mindfulness may sustain decreased symptoms of depression and anxiety at 6-month follow-up, whether it may provide better perceptions of stress and improvement, as well as improving sleep quality, heart rate variability and inflammatory markers at 8-week and, which in turn may enhance response to additional adjunctive therapies (e.g. psychotropic medications), if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18yrs.>
* Currently receiving maintenance hemodialysis, with depression (Patient Health Questionnaire (PHQ-9) score ≥6) and/or anxiety (General Anxiety Disorder-7 (GAD- 7) score ≥6).
* Normal cognition or Mild Cognitive Impairment will be addressed on a normal screening result on the 3-minute Mini-Cog Test (53).
* Patients should have sufficient hearing to follow verbal instructions, be able to sit for 20-25 minutes without discomfort
* Have adequate understanding of English and/or French

Exclusion Criteria:

* Mild, Moderate, or Severe Dementia ("Abnormal" Result on the 3-minute Mini-Cog Test (53))
* Acute psychotic symptoms,
* Acute suicidal ideation/intent
* Patients currently receiving active psychotherapy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Depression scores measured by the Patient Health Questionnaire (PHQ-9) | Baseline, 8 weeks and 6 months
  Represents a self-reported 9-item depression scale and it is based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for major depressive disorder with responses to questions ranging from 0 ("not at all") to 3 ("nearly every day") for each item. Low scores are equivalent to less symptoms of depression (scale range is 0 to 27, 9 items). Summed scores ≥10 are considered clinically significant.
  Our primary endpoint is change in PHQ-9 scores between baseline and 8-weeks. Our primary analysis will be in the subgroup of patients randomized into the study with a baseline PHQ-9 score ≥10. Our secondary analysis for this primary outcome will be with all patients randomized into the study (PHQ-9 or GAD-7 ≥6).

SECONDARY OUTCOMES:
Anxiety scores measured by the General Anxiety Questionnaire (GAD-7) | Baseline, 8 weeks and 6 months
  Represents a self-reported 7-item tool to measure the severity of various signs of generalized anxiety disorder on a 0 ("not at all") to 3 ("nearly every day") scale. Low scores are equivalent to less symptoms of anxiety (scale range is 0 to 21). Summed scores ≥10 are considered clinically significant.
  Our main endpoint for this secondary outcome is change in GAD-7 scores between baseline and 8-weeks. Our primary analysis will be in the subgroup of patients randomized into the study with a baseline GAD-7 score ≥10. Our secondary analysis for this secondary outcome will be with all patients randomized into the study (PHQ-9 or GAD-7 ≥6).

OTHER OUTCOMES:
Perceived Stress Scale (PSS) | Baseline and 8 weeks
  It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. Scale range is 0 to 40. Interpreting scores: 0-7=very low health concern, 8-11 is a low health concern, 12-15= average health concerns, 16-20=high health concern, 21+ =very high health concern.
Perceived Improvement Questionnaire (PIQ) | At program end (8 weeks)
  The PIQ is a standardized questionnaire evaluating changes perceived by patients while receiving outpatient psychiatric services. The PIQ comprises 20 items, one referring to the patient's general situation at the end of treatment (ranges between -40 and 20). Answers are selected from among: ''worse than before = -1'', ''no change = 0'', ''better than before = 1'', and ''much better than before = 2''. Lower scores indicate less perceived improvement from treatment.
Athens Insomnia Scale (AIS) | Baseline and 8 weeks
  The AIS is a self-administered psychometric instrument consisting of eight items assessing difficulty with sleep induction, awakenings during the night, early morning awakening, total sleep time, overall quality of sleep, and the requirements of a minimum frequency (at least three times a week) and duration (1 month) of any complaint. Each item of the AIS can be rated 0 ±3, (with 0 corresponding to ''no problem at all'' and 3'' very serious problem''). The respondents are requested to rate positive if they had experienced the sleep difficulty described in each item at least three times a week during the last month or some other period of time, whose length depends on the purpose of a given study. Total score ranging from 0 (denoting absence of any sleep-related problem) to 24 (representing the most severe degree of insomnia).
Patient's assessment on Quality of Life (EuroQOL) | Baseline and 8 weeks
  It provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys. The EuroQOL essentially consists of 2 pages - the descriptive system and the visual analogue scale (VAS).The EuroQOL descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems.The VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. For descriptive profile, lower scores indicate increased quality of life and for the VAS, higher scores indicate greater overall health.
Edmonton Symptom Assessment Scale (ESAS) | Baseline and 8 weeks
  Developed to assist in the assessment of nine symptoms that are common in palliative care patients: pain, tiredness, drowsiness, nausea, lack of appetite, depression, anxiety, shortness of breath, and well being. The severity at the time of assessment of each symptom is rated from 0 to 10 on a numerical scale, 0 meaning that the symptom is absent and 10 that it is of the worst possible severity. Consists of 9 items (score range 0-90) Lower scores indicate less severity.
Social Difficulties Inventory (SDI) | Baseline and 8 weeks
  DI-21 as part of the assessment guidance for the social and occupational domain of Holistic Common Assessment of Supportive and Palliative Care Needs for Adults with Cancer. The scoring ranges from no diﬃculty to very much diﬃculty (0-3). Consists of 21 items (score range 0-63). Lower scores indicate less difficulty.
Inflammatory markers (blood draw) | Baseline and 8 weeks
  Patients undergoing dialysis also often have a high burden of systemic inflammation, including elevated blood inflammation biomarkers. This in turn triggers a cascade that has been extensively shown in humans and animals to cause depressive symptoms, due to the permeability of blood endothelial cells, followed by activation of inflammatory pathways in the brain (28442354) and consequently, symptoms of depression. A possible association between these pro-inflammatory cytokines and the symptoms of depression can better explain the high rates of depression and the non-adherence to treatment in patients undergoing dialysis.
Heart rate variability (HRV) | Baseline and 8 weeks
  Heart Rate Variability Logger (an IPhone validated application to measure HRV) lets you record, plot and export time and frequency domain Heart Rate Variability Features (includes experience sampling, rr-interval correction, comparison between recordings, activity monitoring & step counting, location tracking).
Circadian rhythm and sleep quality | Baseline and 8 weeks
  Calculation of a mean for absolute time and variation (standard deviation) of sleep onset, sleep offset, duration of sleep, and total inactivity in 24 hours during the study period to describe regularity and timing of sleep. Participants will wear and ActiWatch as a measure of actigraphy for a period of two weeks previous and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Soham Rej, MD/MSc, Principal Investigator — Psychiatrist and researcher
Locations (2):
- Canada (2):
  - Lady David Institute, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Thomas Z, Novak M, Platas SGT, Gautier M, Holgin AP, Fox R, Segal M, Looper KJ, Lipman M, Selchen S, Mucsi I, Herrmann N, Rej S. Brief Mindfulness Meditation for Depression and Anxiety Symptoms in Patients Undergoing Hemodialysis: A Pilot Feasibility Study. Clin J Am Soc Nephrol. 2017 Dec 7;12(12):2008-2015. doi: 10.2215/CJN.03900417. Epub 2017 Oct 12. PMID 29025788
- [Derived] Rigas C, Park H, Nassim M, Su CL, Greenway K, Lipman M, McVeigh C, Novak M, Trinh E, Alam A, Suri RS, Mucsi I, Torres-Platas SG, Noble H, Sekhon H, Rej S, Lifshitz M. Long-term Effects of a Brief Mindfulness Intervention Versus a Health Enhancement Program for Treating Depression and Anxiety in Patients Undergoing Hemodialysis: A Randomized Controlled Trial. Can J Kidney Health Dis. 2022 Mar 4;9:20543581221074562. doi: 10.1177/20543581221074562. eCollection 2022. PMID 35273807
- See also: Related Info — http://geriparty.com